CLINICAL TRIAL: NCT03555422
Title: A Randomized, Double-Blind, Phase 3 Trial of Maintenance with Selinexor/ Placebo After Combination Chemotherapy for Patients with Advanced or Recurrent Endometrial Cancer
Brief Title: Maintenance with Selinexor/Placebo After Combination Chemotherapy in Participants with Endometrial Cancer [SIENDO]
Acronym: ENGOT-EN5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Collaborators: Belgian Gynaecological Oncology Group (Other); North-Eastern German Society of Gynaecologic Oncology (Unknown); Multicentre Italian Trials in Ovarian Cancer and Gynecologic Malignancies (Unknown); Spanish Research Group in Ovarian Cancer (Unknown); The Central and Eastern European Gynecologic Oncology Group (Other); Israeli Society of Gynecologic Oncology (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KCP-330-024; ENGOT-EN5 (Other: European Network of Gynaecological Oncological Trial Groups); BGOG-EN5 (Other: Belgium and Luxembourg Gynaecological Oncology Group); 2017-000607-25 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Neoplasms; Uterine Neoplasms; Genital Neoplasms; Neoplasms by Site; Neoplasms; Uterine Diseases; Genital Diseases; Female
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Neoplasms by Site; Neoplasms; Uterine Diseases; Genital Diseases | interventions — selinexor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind placebo controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selinexor (Experimental): Participants will receive fixed dose of selinexor 80 mg (or 60 mg for participants with a body mass index [BMI] less than [<] 20 kilogram per meter square [kg/m^2]) oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: Selinexor
- Matching placebo for selinexor (Placebo Comparator): Participants will receive matching placebo for selinexor oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: Matching placebo for selinexor

INTERVENTIONS:
Drug: Selinexor — Dose: 80 mg (4 tablets) or 60 mg (3 tablets); Dosage form: film-coated, immediate-release tablet of 20 mg each; Route of administration: oral
  Arms: Selinexor
Drug: Matching placebo for selinexor — Dose: 80 mg (4 tablets) or 60 mg (3 tablets); Dosage form: film-coated, immediate-release tablet of 20 mg each; Route of administration: oral
  Arms: Matching placebo for selinexor

SUMMARY:
This is a prospective, multicenter, double-blind, placebo-controlled, randomized Phase 3 study. The purpose of the study is to obtain evidence of efficacy for maintenance selinexor in participants with advanced or recurrent endometrial cancer. Participants with primary stage IV or recurrent disease who are in partial or complete response after having completed a single line of at least 12 weeks of taxane-platinum combo therapy will be randomized in a 2:1 manner to maintenance therapy with 80 milligram (mg) with selinexor once weekly (QW) or placebo until progression.

ELIGIBILITY:
Inclusion Criteria:

* Female, at least 18 years of age at the time of informed consent.
* Histological confirmed endometrial cancer of the endometrioid, serous, or undifferentiated type. Carcinosarcoma of the uterus is also allowed.
* Completed a single line of at least 12 weeks of taxane-platinum combination therapy (not including adjuvant or neoadjuvant therapy), and achieved partial remission (PR) or complete remission (CR) according to RECIST version 1.1 for:
* Primary Stage IV disease, defined as:
* had a primary or later debulking surgery during first-line taxane-platinum therapy with R0 resection (R0 resection indicates a macroscopic complete resection of all visible tumor) and achieved CR after at least 12 weeks taxane-platinum chemotherapy, OR
* had a primary or later debulking surgery during first-line taxane-platinum therapy with R1 resection (R1 resection indicates incomplete removal of all macroscopic disease,) and achieved PR or CR after at least 12 weeks taxane-platinum chemotherapy, OR
* had no surgery and achieved PR or CR after at least 12 weeks taxane-platinum chemotherapy.

OR

* At first relapse (i.e., relapse after primary therapy including surgery and/or chemotherapy therapy for Stage I-IV disease), defined as:
* had Stage I-III disease at diagnosis and received at initial diagnosis adjuvant chemotherapy and relapsed later. Participants should have PR or CR after at least 12 weeks of taxane-platinum chemotherapy compared with the start of this chemotherapy at the time of relapse, OR
* had Stage I-III disease at diagnosis and did not receive adjuvant chemotherapy at initial diagnosis and relapsed later. Participants should have PR or CR after at least 12 weeks of taxane-platinum chemotherapy compared with the start of this chemotherapy at the time of relapse, OR
* had Stage IV disease at diagnosis and received initially chemotherapy with or without surgery and relapsed later. At the time of relapse, participants should have PR or CR after at least 12 weeks of taxane-platinum chemotherapy compared with the start of this chemotherapy at the time of relapse.

Participants that required their chemotherapy dose held during the 12-week therapy may be considered if they meet the other criteria above and achieve PR or CR per RECIST V1.1.

* Must be able to initiate study drug 5 to 8 weeks after completion of their final dose of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Participants must have adequate bone marrow function and organ function within 2 weeks before starting study drug as defined by the following laboratory criteria:
* Hepatic function: total bilirubin up to 1.5*upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to (≤) 2.5*ULN in participants without liver metastasis. For participants with known liver involvement of their tumor: AST and ALT ≤5*ULN.
* Hematopoetic function: Absolute neutrophil count (ANC) greater than or equal to (≥) 1.5*10^9/L; platelet count ≥100*10^9 per liter (/L); hemoglobin ≥9.0 gram per deciliter (g/dL).
* Renal function: estimated creatinine clearance (CrCl) of ≥20 milliliter per minute (mL/min), calculated using the Cockroft Gault formula.
* In the opinion of the Investigator, the participant must:
* Have a life expectancy of at least 12 weeks, and
* Be fit to receive experimental therapy.
* Premenopausal females of childbearing potential must have a negative pregnancy test (serum β-human chorionic gonadotropin test) prior to the first dose of study drug. Female participants of childbearing potential must agree to use highly effective methods of contraception throughout the study and for 1 week following the last dose of study drug.
* Written informed consent in accordance with federal, local, and institutional guidelines. The participant must provide informed consent prior to the first Screening procedure.

Exclusion Criteria:

* Has any sarcomas, small cell carcinoma with neuroendocrine differentiation, or clear cell carcinomas.
* Received a blood or platelet transfusion during 4 weeks prior to randomization.
* Being treated with a concurrent cancer therapy.
* Previous treatment with an exportin 1 (XPO1) inhibitor.
* Previous treatment with anti- programmed cell death protein 1 (PD-1) or anti-programmed cell death ligand-1 (PD-L1) immunotherapy (e.g., pembrolizumab).
* Concurrent treatment with an investigational agent or participation in another clinical trial.
* Participants who received any systemic anticancer therapy including investigational agents or radiation ≤3 weeks (or ≤5 half-lives of the drug [whichever is shorter]) prior to cycle 1 day 1 (C1D1). Palliative radiotherapy may be permitted for symptomatic control of pain from bone metastases in extremities, provided that the radiotherapy does not involve target lesions, and the reason for the radiotherapy does not reflect progressive disease (PD).
* Major injuries or surgery within 14 days prior to C1D1 and/or planned surgery during the on-treatment study period.
* Previous malignant disease, except participants with other malignant disease, for which the participant has been disease-free for at least 3 years. Concurrent other malignant disease except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin.
* Any life-threatening illness, medical condition or organ system dysfunction, which, in the investigator's opinion, could compromise the participant's safety or compliance with the protocol.
* Known contraindications to selinexor.
* Known uncontrolled hypersensitivity to the investigational drug, or to its excipients.
* Radiotherapy to the target lesion within the past 3 months prior to baseline imaging.
* Persistent Grade 3 or 4 toxicity from previous chemotherapy and/or radiotherapy, with the exception of alopecia.
* Active brain metastases (e.g., stable for <8 weeks, no adequate previous treatment with radiotherapy and/or surgery, symptomatic, requiring treatment with anti-convulsants. Corticoid therapy is allowed if administered as stable dose for at least 1 month before randomization).
* Known unstable cardiovascular function:
* Symptomatic ischemia, or
* Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmia are excluded; 1st degree atrioventricular block or asymptomatic left anterior fascicular block /right bundle branch block will not be excluded), or
* Congestive heart failure of New York Heart Association Class ≥3, or
* Myocardial infarction within 3 months
* Females who are pregnant or actively breastfeeding.
* Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to first dose; however, prophylactic use of these agents is acceptable even if parenteral.
* Active hepatitis C and/or B infection.
* Participants unable to swallow tablets, participants with malabsorption syndrome, or any other gastrointestinal (GI) disease or GI dysfunction that could interfere with absorption of study drug. A history of bowel obstruction requiring a nasogastric tube or intravenous infusion during the past 2 months is not allowed (except when this obstruction is caused by surgery or other non-malignant causes).
* Psychiatric illness or substance use that would prevent the participant from giving informed consent or being compliant with the study procedures.
* Participants unwilling or unable to comply with the protocol.
* Persons who have been committed to an institution by official or judicial order.
* Participants with dependency on the Sponsor, Investigator or study site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 263 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Time from randomization until disease progression (PD) or death, whichever occurs first (approximately 12 months after the last participant enrolled)
  Compare progression free survival of the two treatment arms as assessed by the investigator, per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

SECONDARY OUTCOMES:
Progression Free Survival: Assessed by Blinded Independent Central Review (BICR), per RECIST v1.1 | Time from randomization until PD or death, whichever occurs first (approximately 12 months after the last participant enrolled)
  Time from randomization until documented PD or death due to any cause, whichever occurs first. Documented PD will be based on BICR assessments.
Disease Specific Survival (DSS) | Time from randomization until death from endometrial cancer (approximately 12 months after the last participant enrolled)
  Time from randomization until date of death from endometrial cancer.
Overall Survival (OS) | Time from randomization until death (approximately 12 months after the last participant enrolled)
  Time from randomization until date of death from any cause.
Time to First Subsequent Treatment (TFST) | Time from randomization until first therapy initiation after discontinuation of study drug or death, whichever occurs first (approximately 12 months after the last participant enrolled)
  Time from randomization until date of initiation of first therapy after discontinuation of study drug or death, whichever occurs first.
Progression-free Survival After Subsequent Treatment (PFS2) | Time from randomization until second documented PD or death (approximately 12 months after the last participant enrolled)
  Time from randomization until the second documented disease progression or death due to any cause by any cause on any subsequent line of anticancer therapy.
Time to Second Subsequent Treatment (TSST) | Time from randomization until second therapy initiation after discontinuation of study drug or death, whichever occurs first (approximately 12 months after the last participant enrolled)
  Time from randomization until date of initiation of second therapy after discontinuation of study drug or death, whichever occurs first.
Disease Control Rate (DCR) | Time from randomization up to approximately 16 weeks
  Best response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) among patients with PR as best response to prior chemotherapy.
Health-Related Quality of Life (HR-QoL): Measured by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Every 12 weeks during study period, at PD and post PD at 3 and 6 months (approximately 12 months after the last participant enrolled)
  Patient-reported outcomes will be measured by the EORTC QLQ C30 questionnaire.
Health-Related Quality of Life: Measured by EORTC QLQ-EN24 | Every 12 weeks during study period, at PD and post PD at 3 and 6 months (approximately 12 months after the last participant enrolled)
  Patient-reported outcomes will be measured by the EORTC QLQ-EN24 questionnaire.
Health-Related Quality of Life: Measured by EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | Every 12 weeks during study period, at PD and post PD at 3 and 6 months (approximately 12 months after the last participant enrolled)
  Patient-reported outcomes will be measured by the EORTC EQ-5D-5L.
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Occurrence, Nature, and Severity of AEs | From first drug administration up to 30 days after last dose (approximately 12 months after the last patient enrolled)
Number of Participants with Significant Physical Examination, Clinical Laboratory, and Vital Signs Results | From first drug administration up to 30 days after last dose (approximately 12 months after the last patient enrolled)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (19):
  - Arizona Oncology, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists (Sarah Cannon Research Institute), West Palm Beach, Florida
  - Gynecological Cancer Institute of Chicago, Oak Lawn, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - HCA Midwest Health - Kansas City (Sarah Cannon Research Institute), Kansas City, Missouri
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma Health Sciences Center - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Tennessee Oncology Nashville (Sarah Cannon Research Institute), Nashville, Tennessee
  - Texas Oncology, Austin, Austin, Texas
  - Texas Oncology DFW, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology DFW, Fort Worth, Texas
  - VCU Massey Cancer Center, Richmond, Virginia
- Belgium (6):
  - UZ Gent, Ghent
  - Jan Yperman Ziekenhuis, Ieper
  - Universitaire Ziekenhuizen K.U. Leuven, Leuven
  - CHU UCL Namur, Site Sainte-Elisabeth, Namur
  - AZ Turnhout, Turnhout
  - CHR Verviers, Verviers
- Canada (3):
  - London Health Sciences Centre (London Regional Cancer Centre), London, Ontario
  - University Health Network (PMCC), Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- China (8):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Chongqing University Cancer Hospital, Chongqing, Shapingba District
  - Wenzhou Medical University - The First Affiliated Hospital, Wenzhou, Zhejiang
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Ostrava, Ostrava
  - UH Královské Vinohrady, Prague
  - General University Hospital in Prague, Prague
  - Hospital Na Bulovce, Prague
- Germany (8):
  - Charite Berlin Universitatsmedizin, Berlin
  - University Hospital Dresden, Dresden
  - DIAKOVERE KH gGmbH, Henriettenstift Hannover, Hanover
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitätsfrauenklinik Mainz, Mainz
  - Klinikum der Universitat Munchen, Munich
  - Cartitas Klinikum Saarbrücken, Saarbrücken
  - Universitätsfrauenklinik Ulm, Ulm
- Greece (3):
  - Iaso Hospital, Marousi, Athens
  - ALEXANDRA Hospital, Athens, Greece
  - Euromedica General Clinic, Thessaloniki, Macedonia
- Israel (5):
  - Hillel Yaffe Medical Center, Hadera
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (7):
  - Istituto di Candiolo, FPO, IRCCS, Candiolo
  - Romagnolo Scientific Institute for the Study and Treatment of Tumors, Meldola
  - San Raffaele Hospital, Milan
  - Istituto Nazionale dei Tumori IRCCS - MILANO S.C. Ginecologia Oncologica, Milan
  - ULSS 3 SERENISSIMA UOC Oncologia Ed Ematologia Oncologica, Mirano
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale" - NAPOLI Struttura Complessa Oncologia Medica Uro-Ginecologica, Naples
  - Agostino Gemelli University Polyclinic Foundation, Rome
- Spain (14):
  - Hospital Universitario Donostia, San Sebastián, Gipuzkoa
  - Hospital Universitari Vall d' Hebrón, Barcelona
  - Hospital Universitari Clínic de Barcelona, Barcelona
  - Consorci Sanitari de Terrassa, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Virgen de la Arrixaca University Clinical Hospital, Murcia
  - Hospital Son Llàtzer, Palma
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vergote I, Perez-Fidalgo JA, Hamilton EP, Valabrega G, Van Gorp T, Sehouli J, Cibula D, Levy T, Welch S, Richardson DL, Guerra EM, Scambia G, Henry S, Wimberger P, Miller DS, Klat J, Martinez-Garcia J, Raspagliesi F, Pothuri B, Romero I, Bergamini A, Slomovitz B, Schochter F, Hogdall E, Farinas-Madrid L, Monk BJ, Michel D, Kauffman MG, Shacham S, Mirza MR, Makker V; ENGOT-EN5/GOG-3055/SIENDO Investigators. Oral Selinexor as Maintenance Therapy After First-Line Chemotherapy for Advanced or Recurrent Endometrial Cancer. J Clin Oncol. 2023 Dec 10;41(35):5400-5410. doi: 10.1200/JCO.22.02906. Epub 2023 Sep 5. PMID 37669480